CLINICAL TRIAL: NCT04550689
Title: A Pilot RCT Study Comparing Dimensional Alterations After Socket Grafting With Xenograft Versus Allograft
Brief Title: Comparison of Dimensional Changes After Tooth Extractions Between Xenograft and Allograft
Acronym: PilotXenAllo
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Sejal Thacker, D.D.S., M.D.Sc., Graduate Program Director, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-137-1; 601907 (Other Grant/Funding Number: Straumann LLC)
Record Dates: First submitted 2020-09-07; First posted 2020-09-16 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Tooth Loss
Keywords: dental; socket grafting; bone graft; alveolar; xenograft; allograft; implant; ridge preservation; CBCT
MeSH Terms: conditions — Tooth Loss | interventions — Bone Transplantation

STUDY DESIGN:
Intervention Model Description: Parallel arm with subjects randomly receiving allograft or xenograft for ridge preservation
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participant, surgeon and assessors of the CBCT will be blinded to the treatment arm. The bone graft will be chosen at random from an envelope with a list generated by Sealed Envelope Ltd
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Xenograft (Active Comparator)
  Interventions: Device: Bone graft
- Allograft (Active Comparator)
  Interventions: Device: Bone graft

INTERVENTIONS:
Device: Bone graft — Bone grafts produced by Straumann LLC

SUMMARY:
To compare dimensional changes in extraction socket of single rooted teeth, 6 months post extraction, when grafted with xenograft versus allograft.

DETAILED DESCRIPTION:
AIM To compare dimensional changes in extraction socket of single rooted teeth, 6 months post extraction, when grafted with xenograft versus allograft.

PRIMARY OBJECTIVE

Horizontal and vertical dimensional changes of extraction sockets as evaluated in a CBCT scan immediately post extraction and 6 months post extraction when grafted with xenograft versus allograft.

SECONDARY OBJECTIVE

1. Difference in horizontal dimensional changes in xenograft and allograft groups as measured intra-operatively after extraction and at re- entry 6 months post extraction.
2. Difference in vertical dimensional changes in xenograft and allograft groups as measured intra-operatively after extraction and at re- entry 6 months post extraction.
3. Difference in histologic analysis of bone biopsy cores taken in xenograft and allograft groups at 6 months re-entry from osteotomy site.

Difference in newly regenerated supracrestal bone height and volume will be measured directly from the segmented images from MicroCT.

NULL HYPOTHESIS

There is no difference between the two groups for any of the parameters evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 21 years of age
2. Able to provide informed consent
3. Good general oral health (no active periodontal disease, absence of hopeless teeth, absence of active caries, absence of acute infections)
4. Single rooted non molar teeth needing extraction for miscellaneous reasons (since histological analysis is being done, it is essential to harvest bone core biopsies without inclusion of native bone16)
5. Presence of natural teeth adjacent to the tooth planned for extraction
6. Absence of acute signs of infection such as pus discharge, fistulous tract and / or abscess in relation to tooth being extracted
7. Dehiscence type defects of the sockets limited to 2/3rd length of the root

Exclusion Criteria:

Systemic conditions

1. Conditions and circumstances as evaluated by investigator that would prevent completion of study participation
2. Conditions requiring chronic routine use of antibiotics or steroids
3. History of leukocyte dysfunction or deficiencies, bleeding disorders, neoplastic disease requiring radiation or chemotherapy, metabolic bone disorder, uncontrolled endocrine disorders, HIV infections
4. Alcoholism or drug abuse and heavy smokers >10 cigarettes a day
5. Simultaneous participation in other studies
6. Pregnancy - Patients pregnant before the start of the study or patients who become pregnant during the course of the study

Local conditions

1. Untreated periodontitis, caries or presence of hopeless teeth (other than the one planned for extraction)
2. Multi rooted teeth
3. Irradiation therapy
4. Osseous lesions
5. Missing teeth adjacent to the tooth being extracted
6. Implant restorations adjacent to the tooth being extracted
7. Multiple socket walls missing following extraction or buccal dehiscence defect extending to the apex of the root

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Horizontal and vertical dimensional changes noted on Cone Beam Computed Tomography | 6 months
  Dimensional changes measured from a Cone Beam Computed Tomography immediately post extraction and grafting and 6 months post extraction

SECONDARY OUTCOMES:
Horizontal dimensional changes measured intra-operatively using a Periodontal Probe | 6 months
  Dimensional changes of the crest measured intra-operatively immediately post extraction and grafting and compared to 6 months post extraction. Measurements will be made using a periodontal probe from the Mid-buccal to the mid-palatal/mid-lingual aspect of the ridge using a surgical stent
Vertical dimensional changes measured intra-operatively using a periodontal probe and stent | 6 months
  Dimensional changes of the crest measured intra-operatively immediately post extraction and grafting and compared to 6 months post extraction. Vertical measurements will be made using a periodontal probe and a patient specific stent. The probe will help measure changes in height of buccal and palatal / lingual plate at the center of the ridge.
Histologic analysis of bone biopsy cores | 6 months
  Histologic analysis of the bone biopsy cores taken from the xenograft or allograft grafted extraction sockets

CONTACTS AND LOCATIONS:
Overall Officials: Sejal Thacker, D.D.S., Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No